CLINICAL TRIAL: NCT02298894
Title: Comparison of LDL-P With LDLC From VAPII, NMR, and Ion Mobility
Brief Title: Comparison of LDL Particle Count With Other Available Lipid Tests
Acronym: LIPID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Scripps Clinic (Other)
Responsible Party: Sponsor
Organization: Scripps Health (Other)
Other Study IDs: SCIML001
Record Dates: First submitted 2014-10-27; First posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-10

CONDITIONS: Hyperlipidemia
Keywords: Low Density Lipoprotein (LDL); Lipoprotein; Nuclear Magnetic Resonance (NMR); Vertical Auto Profile (VAP); Ion mobility; Apoliproprotein B (ApoB)
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum, and plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Despite the wide availability of advanced lipoprotein tests, no reference standard exists for Low Density Lipoprotein Cholesterol (LDL-C) due to inherent problems with each of the assays. Newer methods for estimating LDL particle numbers, including nuclear magnetic resonance (NMR) spectroscopy and vertical auto profile (VAP) are currently under investigation. NMR has been proposed as having the best correlation with adverse cardiovascular outcomes. Unfortunately, the accuracy of LDL-C or LDL particle number measurements is currently not monitored by national standardization programs. Direct comparisons between the various testing methods have been limited restricting our ability to accurately interpret and compare values across vendors and lipid parameters.

Our hypothesis is that:

1. LDL particle count numbers, as determined by NMR (Liposcience), provides the best estimates of cardiovascular risk.
2. Discrepancies exist between the LDL particle count by NMR and other values as presented by calculated LDLC and directly measured LDL (VAP and ion mobility).

The investigators will enroll 100 patients recruited from the Lipid Clinic at the Scripps Center for Integrative Medicine. Each patient will have one blood draw from which four tests will be analyzed. Risks are associated with drawing blood, which will be minimized by using Scripps Clinic Lab technicians. The potential loss of personal health information will be reduced by limiting access to study and lab staff and keeping information password-protected on Scripps servers.

DETAILED DESCRIPTION:
Introduction Advanced lipoprotein testing has been available for over 50 years and its use in cardiovascular risk stratification has been proposed in a number of clinical trials (Superko 2009, 2383). Low Density Lipid Cholesterol (LDLC) is currently used as the key cardiovascular biomarker for assessing risk and monitoring response to lipid therapy (Cole, T. 2013, 752). The highest correlation with cardiovascular risk has been found with apolipoproteinB (apoB) or LDL particle concentration by NMR (Brunzell 2008, 814). Despite the wide availability of advanced lipoprotein tests, no reference standard exists for LDLC due to inherent problems with each of the assays (Mora 2009, 2402)(Marcovina 2006, 440). The most common laboratory method of determining LDLC is by precipitation of apolipoproteinB (apoB) containing lipoprotein particles, measurement of the high density lipoprotein cholesterol (HDLC), and calculation of the LDLC by the Friedewald equation; however, there are inherent errors associated with three separate measurements (Marcovina 2006, Superko 2009, 2384). Correlation between lab LDLC and values obtained by ultracentrifugation has been reported to range from 7 to 31.2%, with a significant amount of misclassification (Marcovina, S. and Packard, C. 2006, 440). Furthermore, elevated triglycerides have been reported to interfere with the accuracy of LDLC measurements (Marcovina, S. and Packard, C. 2006, 440). ApoB, which is the main protein component of LDL, is also considered a direct measure of LDL particle number (Cole, T. 2013, 753). Newer methods for estimating LDL particle number, including NMR and VAP are currently under investigation. NMR has been proposed as having the best correlation with adverse cardiovascular outcomes (reference). Unfortunately, the accuracy of LDLC or LDL particle number measurements is currently not monitored by national standardization programs. Direct comparisons between the various testing methods have been limited limiting our ability to accurately interpret and compare values across vendors and lipid parameters.

Hypothesis:

* LDL particle count numbers determined by NMR (Liposcience) provides the best estimates of cardiovascular risk
* Discrepancies exist between the LDL particle count by NMR and other values:

  * Calculated LDLC
  * Directly measured LDL (VAP and ion mobility)

Objective:

* To determine the test which has the highest concordance and lowest concordance with the NMR test Study Design
* Prospective analysis with a target study population of 100 patients
* Superiority study aimed to detect a 300 point difference in LDL particle count
* Requires a one-time lab draw for all patients

Inclusion criteria

* Greater than 18 years of age
* On statin, statin and natural supplements, or natural supplements only

Exclusion criteria

* Within 6 months from an acute myocardial infarction (MI) or acute coronary syndrome (ACS)
* Non-English speaker

Risks to the patient:

* Loss of personal health information
* Phlebotomy related risks, including injury, bruising, and vasovagal reactions

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age of older
* Can read and write English

Exclusion Criteria:

* Acute coronary syndrome within 6 months from the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are seen in the outpatient setting
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-07 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Comparing the Nuclear Magnetic Resonance (NMR) Low Density Lipid (LDL) particle count with LDL values obtained from other methodologies. | Analysis of values will be completed no later than 3 months after enrollment closes.
  Bland Altman plot describing the correlation between LDL particle count number as measured by NMR in comparison to measurements by VAPII, ion mobility, and ApoB liproprotein precipitation will be determined. The specific unit of measurement will be the actual numbers for each LDL particle.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Triffon, MD, Principal Investigator — Scripps Center for Integrative Medicine
Locations (1):
- Scripps Center for Integrative Medicine, La Jolla, California, United States